CLINICAL TRIAL: NCT06653907
Title: Randomized Control Study of Levothyroxine Intervention in Pregnant Women with Thyroid Stimulating Hormone Between 2.5 MIU/L and Upper Limit of Reference Range and Negative Thyroid Peroxidase Antibody
Brief Title: Levothyroxine Intervention in Pregnant Women with TSH （2.5 MIU/L-upper Limit of Reference Range） and Negative Thyroid Peroxidase Antibody
Acronym: LIGHT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yang ZHANG (Other)
Collaborators: National Research Institute for Family Planning, China (Other Government); The Fourth Hospital of Shijiazhuang (Other)
Responsible Party: Sponsor-Investigator, Yang ZHANG, Associated chief of the endocrinology department of peking university first hospital, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20230099; 2021CR29 (Other Grant/Funding Number: Peking university first hospital)
Record Dates: First submitted 2024-10-14; First posted 2024-10-22 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Thyroid Abnormalities; Pregnant Woman; Pregnancy Outcomes
Keywords: TSH; TPOAb; pregnant women; levothyroxine; outcome
MeSH Terms: conditions — Thyroid Diseases | interventions — Thyroxine; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): The target participants are women who undergo thyroid function and TPOAb testing in early pregnancy. Among these pregnant women, TSH 2.5mIU/L-ULRR and TPOAb negative pregnant women will be selected. Then, participants were randomly assigned 1:1 (based on age and BMI) to an oral placebo group during pregnancy. Participants in our study will determine the dosage of medication based on their weight.
  Interventions: Drug: Placebo
- Levothyroxine (Active Comparator): The target participants are women who undergo thyroid function and TPOAb testing in early pregnancy. Among these pregnant women, TSH 2.5mIU/L-ULRR and TPOAb negative pregnant women will be selected. Then, participants were randomly assigned 1:1 (based on age and BMI) to an active comparator group of oral Levothyroxine (L-T4) during pregnancy. Participants in our study will determine the dosage of medication based on their weight.
  Interventions: Drug: Levothyroxine Sodium (LT4) Tablets

INTERVENTIONS:
Drug: Levothyroxine Sodium (LT4) Tablets — Participants in our study will determine the dosage of L-T4 based on their weight (BW):
  1. BW ≥50kg: Starting with a daily dose of 1 tablet;
  2. BW < 50kg: Starting with a daily dose of half a tablet.
  At 12 weeks, 18-20 weeks, 24-26 weeks, and 34-36 weeks of gestation, the serum TSH, FT3, and FT4 will be measured, and investigator will adjust dosage according to TSH:
  1. When TSH > ULRR, the participants will receive L-T4 in addition to their original medication, and additional unplanned follow-up;
  2. When TSH at 2.5mIU/L-ULRR, add 1/4 tablet of medictaion;
  3. When TSH at LLRR -2.5mIU/L, maintain the original dose;
  4. When TSH <LLRR, reduce 1/4 tablets of medictaion.
  5. If TSH continues to be lower than LLRR after discontinuation, investigator will measure FT4, TRAb and other indicators to determine if it is clinical hyperthyroidism. If so, antithyroid drugs will administered according to guidelines. Participants will stop all trial medictaion after delivery.
  Arms: Levothyroxine
Drug: Placebo — Participants in our study will determine the dosage of placebo based on their weight (BW):
  1. BW ≥50kg: Starting with a daily dose of 1 tablet;
  2. BW < 50kg: Starting with a daily dose of half a tablet.
  At 12 weeks, 18-20 weeks, 24-26 weeks, and 34-36 weeks of gestation, the serum TSH, FT3, and FT4 will be measured, and investigator will adjust dosage according to TSH:
  1. When TSH > ULRR, the participants will receive L-T4 in addition to their original medication, and additional unplanned follow-up;
  2. When TSH at 2.5mIU/L-ULRR, add 1/4 tablet of medictaion;
  3. When TSH at LLRR -2.5mIU/L, maintain the original dose;
  4. When TSH <LLRR, reduce 1/4 tablets of medictaion.
  5. If TSH continues to be lower than LLRR after discontinuation, investigator will measure FT4, TRAb and other indicators to determine if it is clinical hyperthyroidism. If so, antithyroid drugs will administered according to guidelines. Participants will stop all trial medictaion after delivery.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if levothyroxine (L-T4) works to treat pregnant women with TSH 2.5 mIU/L-the upper limit of reference range (ULRR) of pregnancy and TPOAb-negative. It will also learn about the safety of L-T4. The main quesitons the investigator want to answer are:

* Will L-T4 reduce miscarriage rates and have an impact on pregnancy complications in pregnant participants?
* What medical issues do participants have when taking L-T4 during pregnancy? -Investigators will compare L-T4 with placebo (a substance with a similar appearance without medication) to see if L-T4 could reduce miscarriage rates

Participants should:

* Take L-T4 or placebo during the whole pregnancy.
* Visit the hospital once every 6-8 weeks during pregnancy for checkups and tests
* Keep a diary of their pregncny complications and daily record of L-T4 or placebo intake.
* Visit the hospital for examination 42 days postpartum for checkups and follow up by phone at 6 and 12 months postpartum.

ELIGIBILITY:
Inclusion Criteria:

1. Women of childbearing age（18-45 years old）, natural pregnancy, singleton pregnancy.
2. Measure thyroid related indexes within 8 weeks of pregnancy: TSH 2.5mIU/L-ULRR, FT4 is normal and TPOAb negativity.
3. Willing to sign an informed consent form.

Exclusion Criteria:

1. History of recurrent miscarriage (≥3 times).
2. Assisted reproduction (artificial insemination, in vitro fertilization and embryo transfer);
3. Suffer from diseases that seriously affect pregnancy outcome, including hypertension, diabetes, heart disease, liver and kidney dysfunction, etc.
4. Failure of vital organs.
5. Except autoimmune thyroid disease，suffer from other autoimmune diseases.
6. Thyroid diseases (including hyperthyroidism, thyroid cancer, thyroid amyloidosis and other extensive intrathyroidal diseases, current subacute thyroiditis, iodine-deficiency endemic goiter, thyroidectomy or 131I treatment, previous thyroid Ultrasound prompts diffuse thyroid disease, etc.).
7. Use of thyroid-related drugs (lithium carbonate, thioureas, sulfonamides, sodium para-amino salicylate, potassium perchlorate, phenylbutazone, sulfate, tyrosine kinase inhibitor, etc.) during screening and affect thyroid Functional testing drugs. (Including glucocorticoids, metoclopramide, propranolol, amiodarone, sodium valproate, etc.)
8. Secondary hypothyroidism or central hypothyroidism. (Including pituitary tumors, surgery, radiotherapy, lymphocytic hypophysitis, etc.)
9. L-T4 allergy.
10. Unwilling to sign an informed consent.
11. Other clinicians judged that they are not suitable to participate in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 400 (Estimated)
Dates: Start 2024-10-25 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Rate of fetal loss | From enrollment to the end of treatment at 40 weeks
  * Abortion: Ultrasound examination shows no embryo sac or only empty sac, no fetal heart or bud development.
  * Intrauterine fetal death: Fetal death in utero at 20 weeks or more of pregnancy.
  * Stillbirth: Death at birth over 28 weeks of pregnancy.
  * Neonatal death: Newborns die within 7 days.

SECONDARY OUTCOMES:
Fetal loss rates and reasons within 12 weeks of pregnancy. | From enrollment to the end of treatment at 12 weeks
Fetal loss rates and reasons within 24 weeks of pregnancy. | From enrollment to the end of treatment at 24 weeks
Fetal loss rates and reasons within 28 weeks of pregnancy. | From enrollment to the end of treatment at 28 weeks
Fetal loss rates and reasons within 34 weeks of pregnancy. | From enrollment to the end of treatment at 34 weeks
Rate of cesarean section | From enrollment to the end of treatment at 40 weeks
Gestational week of delivery | From enrollment to the end of treatment at 40 weeks
Number of Participants requiring treatments for preventing miscarriage | From enrollment to the end of treatment at 40 weeks
  Drugs, cervical cerclage, etc.
Rate of hyperemesis gravidarum | From enrollment to the end of treatment at 40 weeks
Rate of gestational diabetes | From enrollment to the end of treatment at 40 weeks
  GDM:
  1. FPG≥5.1mmol/L,<7.0mmol/L during the first prenatal examination
  2. During weeks 24-28, if blood glucose was elevated in a 75 g oral glucose tolerance test according to the criteria of International Association of the Diabetes and Pregnancy Study Groups; 0 hour ≥5.1 mmol/L, 1 hour ≥10.0 mmol/L, 2 hours ≥8.5 mmol/L Satisfy any of the above criteria to diagnose GDM
Rate of hypertensive disorders of pregnancy | From enrollment to the end of treatment at 40 weeks
  Hypertensive disorders of pregnancy include: hypertension during pregnancy, preeclampsia and eclampsia
Rate of early preterm delivery | From enrollment to the end of treatment at 34 weeks
  28 weeks ≤ gestational week of delivery <34 weeks;
Rate of late preterm delivery | From enrollment to the end of treatment at 37 weeks
  34 weeks ≤ delivery gestational week <37 weeks
Rate of intrauterine growth restriction | From enrollment to the end of treatment at 40 weeks
Rate of abruption of placenta | From enrollment to the end of treatment at 40 weeks
Rate of dystocia | From enrollment to the end of treatment at 40 weeks
  Dystocia: fetus delivery is difficult, requiring assisted delivery or cesarean section
Rate of macrosomia | From enrollment to the end of newborn delivery date.
  Macrosomia: the newborn's birth weight >=4000 g
Rate of low birth weight | From enrollment to the end of newborn delivery date.
  Low birth weight: the newborn's birth weight <2500 g
Incidence of composite adverse outcomes | From enrollment to the end of treatment at 40 weeks
  The occurrence of one or more of these above events (maternal and fetal) was defined as the occurrence of prenatal composite adverse outcomes.

OTHER OUTCOMES:
Adverse events (AEs) | From enrollment to the end of treatment at 40 weeks
  Any unexpected medical occurrence in a subjects administered a pharmaceutical product and which may have no causal relationship with the treatment. An AE can be the aggravation of original symptoms, signs, laboratory abnormalities or newly diagnosed diseases, unfavorable and unintended symptoms, signs, clinically significant laboratory abnormalities, etc.
  The following situations should not be recorded as AEs:
  * Existing conditions found during first visiting
  * Planned hospitalization/surgery
  * Invasive medical and surgical examinations, however, diseases that require these examinations may be adverse events
  * Expected progression of thyroid disease.
  * Existing accompanying diseases or existing symptoms and signs exhibited the expected periodic fluctuations at the time of screening, but did not worsen
Serious adverse events (SAEs) | From enrollment to the end of treatment at 40 weeks
  Defined as any untoward medical position that meets one or more of the following criteria:
  1. Death
  2. Life-threatening
  3. Requires hospitalisation or prolong existing hospitalisation
  4. Results in disability/incapacity
  5. Results in a birth defect.
Thyrotoxicosis | From enrollment to the end of treatment at 40 weeks
  Defined as serum TSH less than the lower limit of the pregnancy-specific reference range (or 0.1 mU/L).

CONTACTS AND LOCATIONS:
Overall Officials: Ying Gao, Professor, Study Chair — Endocrinology Department of Peking University First Hospital
Locations (1):
- Fourth hospital of Shijiazhuang city, Shijiazhuang, Heibei, China

IPD SHARING:
Plan to Share IPD: Yes
the clinical information of the participants and the primary outcome data of the LIGHT study will be shared
Supporting Information: Study Protocol, CSR
Time Frame: IPD will be available half year after the last participants finished the study